CLINICAL TRIAL: NCT00095875
Title: A Randomized Phase III Comparing Sequential Therapy With TPF/Chemoradiation (ST) To Cisplatinum-Based Chemoradiotherapy [PARADIGM TRIAL]
Brief Title: Combination Chemotherapy and Radiation in Treating Patients With Stage III or IV Head and Neck Cancer (Paradigm Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Medical Oncology, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFCI 04-006; P30CA006516 (NIH); CDR0000393548 (Registry Identifier: NCI PDQ); NCT00705068 (obsolete NCT alias)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Cisplatin; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil. Treatment repeats every 21 days for 3 courses. Patients achieving a pathologic complete response at the primary site and a clinical complete response in the neck then receive carboplatin once weekly and undergo concurrent radiotherapy once daily, 5 days a week, for 7 weeks. Patients with a partial response at the primary site (i.e., positive biopsy), stable disease, or radiographic evidence of persistent disease in the neck receive docetaxel once weekly for 4 weeks and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 6 weeks.
  Interventions: Drug: carboplatin; Drug: cisplatin; Drug: docetaxel; Drug: fluorouracil
- Arm II (Experimental): Patients receive cisplatin IV on weeks 1 and 4 and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 6 weeks.
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Paraplatin
  Arms: Arm I
Drug: cisplatin — Given IV
  Other Names: Platinol
Drug: docetaxel — Given IV
  Other Names: Taxotere
  Arms: Arm I
Drug: fluorouracil — Given IV
  Other Names: Efudex
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, cisplatin, fluorouracil, and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells. It is not yet known which regimen of chemotherapy and radiation therapy is most effective in treating head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of chemotherapy and radiation therapy in treating patients who have stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare 3-year survival of patients with previously untreated stage III or IV squamous cell carcinoma of the head and neck treated with induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil followed by radiotherapy and carboplatin or docetaxel vs radiotherapy and cisplatin only.

Secondary

* Compare 2-year progression-free status in patients treated with these regimens.
* Compare 5-year survival of patients treated with these regimens.
* Compare 3- and 5-year progression-free survival of patients treated with these regimens.
* Compare the complete response rate in patients treated with these regimens.
* Compare tumor site-specific survival in patients treated with these regimens.
* Compare functional organ preservation in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Correlate tissue and germline markers with response, local/regional control, and the development of distant metastases in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil. Treatment repeats every 21 days for 3 courses. Patients achieving a pathologic complete response at the primary site and a clinical complete response in the neck then receive carboplatin once weekly and undergo concurrent radiotherapy once daily, 5 days a week, for 7 weeks. Patients with a partial response at the primary site (i.e., positive biopsy), stable disease, or radiographic evidence of persistent disease in the neck receive docetaxel once weekly for 4 weeks and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 6 weeks.
* Arm II: Patients receive cisplatin IV on weeks 1 and 4 and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 6 weeks.

Quality of life is assessed at baseline and then at 3, 12, and 24 months.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 330 patients will be accrued for this study.

ELIGIBILITY:
List of Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck

  * Stage III or IV* disease
  * One of the following primary tumor sites:

    * Oral cavity

      * No mandible invasion
    * Oropharynx
    * Hypopharynx
    * Larynx
  * The following primary tumor sites are excluded:

    * Nasal cavity
    * Paranasal cavity
    * Nasopharynx NOTE: *No evidence of distant metastases by chest x-ray, abdominal ultrasound, or CT scan (for patients with liver function test abnormalities) or bone scan (for patients with local symptoms)
* At least 1 uni- or bi-dimensionally measurable lesion

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 g/dL

Hepatic

* Bilirubin normal
* AST or ALT within eligibility range
* Alkaline phosphatase within eligibility range

Renal

* Creatinine clearance > 60 mL/min

Cardiovascular

* No unstable cardiac disease despite treatment
* No myocardial infarction within the past 6 months

Pulmonary

* No chronic obstructive pulmonary disease, defined as requiring hospitalization for pneumonia or respiratory decompensation within the past year

  * Obstruction caused by the tumor allowed

Neurologic

* No symptomatic peripheral neuropathy > grade 2
* No symptomatic altered hearing > grade 2
* No history of significant neurologic or psychiatric disorders, including dementia or seizures

Other

* No active drug addiction, including alcohol, cocaine, or intravenous drugs within the past 6 months
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, or other cancer curatively treated by surgery alone
* No active, clinically significant, uncontrolled infection
* No autoimmune disease requiring therapy
* No unhealed or clinically active peptic ulcer disease
* No hypercalcemia
* No other serious illness or medical condition
* No involuntary weight loss > 25% of body weight within the past 2 months
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* No prior organ transplantation
* No prior surgery for this cancer

  * Biopsy allowed

Other

* More than 30 days since prior participation in another investigational study
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2004-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert I. Haddad, MD, Study Chair — Dana-Farber Cancer Institute
Locations (15):
- United States (14):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - UMDNJ University Hospital, Newark, New Jersey
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
- Klinikum der J.W. Goethe Universitaet, Frankfurt, Germany

REFERENCES:
- [Result] Haddad R, O'Neill A, Rabinowits G, Tishler R, Khuri F, Adkins D, Clark J, Sarlis N, Lorch J, Beitler JJ, Limaye S, Riley S, Posner M. Induction chemotherapy followed by concurrent chemoradiotherapy (sequential chemoradiotherapy) versus concurrent chemoradiotherapy alone in locally advanced head and neck cancer (PARADIGM): a randomised phase 3 trial. Lancet Oncol. 2013 Mar;14(3):257-64. doi: 10.1016/S1470-2045(13)70011-1. Epub 2013 Feb 13. PMID 23414589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 24, 2004 and December 29, 2008 145 patients were enrolled across 16 sites.
Pre-assignment Details: Patients were randomly assigned in a 1:1 ratio to recieve either induction chemotherapy with 3 cycles of TPF followed by concurrent chemoradiotherapy with either docetaxel or carboplatin or concurrent chemoradiotherapy alone with 2 cycles of bolus cisplatin.
Groups:
- Arm I: Patients receive induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil. Treatment repeats every 21 days for 3 courses. Patients achieving a pathologic complete response at the primary site and a clinical complete response in the neck then receive carboplatin once weekly and undergo concurrent radiotherapy once daily, 5 days a week, for 7 weeks. Patients with a partial response at the primary site (i.e., positive biopsy), stable disease, or radiographic evidence of persistent disease in the neck receive docetaxel once weekly for 4 weeks and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 6 weeks.
  cisplatin : Given IV
  radiation therapy : Patients undergo radiation therapy once or twice daily, 5 days a week, for up to 7 weeks
  carboplatin : Given IV
  fluorouracil : Given IV
  docetaxel : Given IV
- Arm II: Patients receive cisplatin IV on weeks 1 and 4 and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 6 weeks.
  cisplatin : Given IV
  radiation therapy : Patients undergo radiation therapy once or twice daily, 5 days a week, for up to 7 weeks
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 70 | 75
Completed | 56 | 66
Not Completed | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 70 | 75 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 66 | 125
  >=65 years | 11 | 9 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (9) | 54 (8) | 55 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 64 | 63 | 127
Region of Enrollment [Number; unit: participants]
  United States | 69 | 69 | 138
  Germany | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To compare the 3-year survival achieved by docetaxel/cisplatin/5-FU based sequential therapy with platinum based chemo radiotherapy in patients with locally advanced SCCHN. Overall survival is defined as the time from date of randomisation to death from any cause. Patients alive at the time of current analysis were censored at the date last known to be alive.Kaplan-Meier method was used to estimate overall survival
Time Frame: 3-years
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 70 | 75
percent of patients | 73 [60 to 82] | 78 [66 to 86]

2. Secondary Outcome: Progression-free Survival and Disease-specific Survival as Assessed by Disease Progression or Death and Log Rank Tests at the Median, and 2, 3, and 5 Years
Description: Progression free survival was defined as the time from date of randomisation to disease progression or death from any cause without progression whichever occurred first; otherwise, patients were censored at the date last known to be free of progression.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percent of patients
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 70 | 75
percent of patients | 67 [54 to 76] | 69 [56 to 79]

ADVERSE EVENTS:
Description: Only the following adverse events were records: mucositis, febrile neutropenia, pain, xerostomia, feeding tube placement, and neuropathy which was deemed pertinent to the comparision of regimens in this setting.
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 56/70 | 29/75
Other Adverse Events (participants affected / at risk) | 70/70 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=70) | Arm II (N=75)
Mucositis (Gastrointestinal disorders) | 33 | 12
Febrile Neutropenia (Blood and lymphatic system disorders) | 16 | 1
Pain (General disorders) | 2 | 9
Xerostomia (Gastrointestinal disorders) | 5 | 5
Neurpathy (Nervous system disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=70) | Arm II (N=75)
Mucositis (Gastrointestinal disorders) | 29 | 44
Pain (General disorders) | 41 | 35
Xerostomia (Gastrointestinal disorders) | 42 | 46
Neuropathy (Immune system disorders) | 22 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes